CLINICAL TRIAL: NCT05801549
Title: Arterio-Venous Fistula Audit. Successful Utilisation Rates of Arterio-Venous Fistulae for Haemodialysis at University Hospital Limerick
Status: Completed | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, CNM II Research, University Hospital of Limerick
Other Study IDs: DVS007
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Arterio-venous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We wish to examine Arterio-Venous Fistula (AVF) and Arterio-Venous Graft (AVG) utilisation rates for Haemodialysis at University Hospital Limerick. We want to determine out of the AVF's that are surgically created, how many go on to be used as anticipated for haemodialysis treatments successfully.

DETAILED DESCRIPTION:
There are over 2 million end-stage renal disease (ESRD) patients who require renal replacement therapy worldwide, and this is estimated to rise to over 5 million by 2030 (Liyanage et al. 2015).

Haemodialysis, used by the majority of ESRD patients, requires vascular access, where blood can be taken out of the body (via cannulation) and pumped through an external dialysis machine, which filters the blood of waste and excess fluid before being returned.

Arterio-venous fistula creation is the preferred vascular access for haemodialysis, but has a large failure rate in the maturation period (Colley et al. 2022). Failure is usually attributed to insufficient dilation of the vessel and/or stenosis, which results in inadequate blood flow rates for the purpose of haemodialysis (Dixon, 2006).

The purpose of this audit is to examine over a three year period how many of the individuals who had an AVF created are utilising it successfully for the purpose of haemodialysis as planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an AVF or AVG surgically created over the last three years at UHL who are undergoing haemodialysis treatments are suitable for inclusion.
* Dates for audit purposes are 1st April 2019 to 1st April 2022.

Exclusion Criteria:

* Patients outside of these set dates will be excluded.
* Patients who are not currently undergoing haemodialysis treatments are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had an AVF or AVG surgically created over the last three years at UHL who are undergoing haemodialysis treatments are suitable for inclusion.
  Dates for audit purposes are 1st April 2019 to 1st April 2022.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Number of AVF's created | 3 years
  We will determine how many were created surgically during the time frame.

SECONDARY OUTCOMES:
AVF's in use for the purpose of Haemodialysis | 3 years
  We will dtermine how many are in use for haemodialysis as planned.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Colley, E., Carroll, J., Anne, S., Shannon, T., Ramon, V. and Tracie, B. (2022). A longitudinal study of the arterio-venous fistula maturation of a single patient over 15 weeks. Biomechanics and Modeling in Mechanobiology, pp.1-16. Dixon, B.S. (2006). Why don't fistulas mature? Kidney International, 70 (8): pp1413-1422. Liyanage, T., Ninomiya, T., Jha, V., Neal, B., Patrice, H.M., Okpechi, I., Zhao, M.H., Lv, J., Garg, A.X., Knight, J. and Rodgers, A. (2015). Worldwide access to treatment for end-stage kidney disease: a systematic review. The Lancet, 385 (9981), pp.1975-1982.